CLINICAL TRIAL: NCT00773097
Title: Study of the MUC1 Peptide - Poly-ICLC Adjuvant Vaccine in Individuals With Advanced Colorectal Adenoma
Brief Title: Study of the MUC1 Peptide-Poly-ICLC Adjuvant Vaccine in Individuals With Advanced Colorectal Adenoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Schoen (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Schoen, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO07030214
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Risk for Colorectal Cancer
Keywords: Prevention; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MUC1 Poly-ICLC (Experimental)
  Interventions: Biological: MUC1 - Poly ICLC

INTERVENTIONS:
Biological: MUC1 - Poly ICLC — The vaccine will be administered on an outpatient basis in the Digestive Disorders Clinic. The total volume of each dose of vaccine MUC1+ POLY-ICLC will be approximately 250 microliters subcutaneously (SQ) in the upper thigh. The site of injection will remain the same thigh, to enhance the potential immune response.

SUMMARY:
The purpose of this study is to evaluate the immune response to MUC1 - poly-ICLC vaccine, an investigational or study vaccine. The MUC1 - poly-ICLC vaccine is being tested in persons with a history of advanced adenomatous polyps, the precursor to colorectal cancer. The MUC1 - poly-ICLC vaccine is being developed to prevent polyps from advancing into colon cancer and to prevent polyps from recurring.

MUC1 is mucus that is normally present on the lining of the human colon. However, MUC1 is expressed in a larger amount and in a modified form on adenomatous polyps and colorectal cancer. These changes in MUC1 are thought to be part of the process of progression from adenomas toward cancer. The goal of a vaccine is to help the immune system in the body identify the changes in MUC1 that accompany the progression to cancer and eliminate the abnormal cells that make abnormal MUC1.

DETAILED DESCRIPTION:
This is a phase II trial designed to assess antibody and T cell responses to MUC1 vaccine among subjects at increased risk for colorectal cancer by virtue of a history of advanced adenoma. The primary objective is to evaluate the immunogenicity of a combination of the 100mer MUC1 peptide and adjuvant Poly-ICLC in boosting the immune response to MUC1. Among the secondary objectives is to determine if anti-MUC1 immunity, preexisting or vaccine induced, has an effect on the recurrence of polyps. Subjects with a history of advanced adenoma will be recruited for MUC1 vaccination. Vaccine will be administered at weeks 0, 2, and 10. Some subjects may have pre-existing immunity to MUC1, and this will be accounted for in the analytic phase. However, all subjects will be administered the vaccine, regardless of baseline antibody status. To insure accurate standardization in measurement and assessment of antibody levels, assays for baseline antibody status will be done at the same time as those for response to vaccine.

ELIGIBILITY:
Inclusion Criteria:

-Age 40 - 70 years of age.

* History of any of the following conditions (operative notes, endoscopy reports, and/or pathology reports must be reviewed locally to confirm that the candidate meets at least one of the following entry criteria).

  1. Colorectal adenoma(s) ≥ 1 cm in maximal diameter
  2. Colorectal adenoma(s) with villous or tubulovillous histology
  3. Colorectal adenoma(s) with high-grade dysplasia
* Willingness to avoid pregnancy or impregnate (see below) for the period of active study (1 year).
* ECOG performance status 0 or 1
* Hemoglobin greater than 95% of the lower limit of institutional normal. Platelets ≥100,000/µL.
* AST (SGOT), ALT (SGPT), alkaline phosphatase, total bilirubin, BUN, creatinine ≤ 1.5x upper limit of institutional normal.
* ANA < 1:160

Exclusion Criteria:

* Receiving any other investigational agents.
* Presence of an active acute or chronic infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to the study agents.
* History of heritable cancer syndrome (FAP, HNPCC)
* Patients with a history of auto-immune disease such as, but not restricted to, inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, ankylosing spondylitis, scleroderma, or multiple sclerosis.
* History of malignancy < 5 years prior to the Registration/Randomization evaluation, excluding non-melanoma skin cancer.
* Any use of oral corticosteroids ≤ 12 weeks prior to Registration/Randomization.
* Current or planned use of immunomodulators including: Remicade, 6-MP (Mercaptopurine), Methotrexate, cyclosporine, or other immunomodulatory drugs.
* Pregnant women, because the teratogenic or abortifacient effects of the study agents remain incompletely defined. Breastfeeding women, because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with the study agents.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2008-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Schoen, Principal Investigator — University of Pittsburgh
Locations (1):
- Digestive Disorders Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Kimura T, McKolanis JR, Dzubinski LA, Islam K, Potter DM, Salazar AM, Schoen RE, Finn OJ. MUC1 vaccine for individuals with advanced adenoma of the colon: a cancer immunoprevention feasibility study. Cancer Prev Res (Phila). 2013 Jan;6(1):18-26. doi: 10.1158/1940-6207.CAPR-12-0275. Epub 2012 Dec 17. PMID 23248097

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient recruitment took place at the University of Pittsburgh Digestive Disorders Clinic. Start date for enrollment was November 11, 2008 - February 16, 2011
Pre-assignment Details: The subjects were excluded if they had a history of a heritable cancer syndrome, autoimmune disease, or a malignancy within 5 years before the enrollment, excluding nonmelanoma skins cancer.
Groups:
- MUC1 Poly-ICLC: MUC1 - Poly ICLC : The vaccine will be administered on an outpatient basis in the Digestive Disorders Clinic. The total volume of each dose of vaccine MUC1+ POLY-ICLC will be approximately 250 microliters subcutaneously (SQ) in the upper thigh. The site of injection will remain the same thigh, to enhance the potential immune response.
Period: Overall Study
Arm/Group | MUC1 Poly-ICLC
Started | 46
Completed | 39
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Population: A total of 39 subjects completed the 52 weeks of the study.
Arm/Group | MUC1 Poly-ICLC
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti Muc-1 Antibody
Description: Evaluation of the immune response to MUC1 peptide vaccine administered with Poly-ICLC, measured by Anti MUC1 antibody, in patients with a history of advanced colorectal adenoma.
Time Frame: 52 weeks
Population: Of the 46 subjects who consented to participate, 6 did not receive vaccine: 4 had abnormal screening laboratory test, 1 did not meet criteria for an advanced adenoma, and 1 declined to participate
Measure: Number; unit: participants
Arm/Group | MUC1 Poly-ICLC
Number analyzed (Participants) | 39
participants | 39

2. Secondary Outcome: Number of Participants With Autoimmune Response to Muc-1 Vaccine
Description: Evaluate for autoimmune response by measuring the Anti-muc-1 IgG antibodies to the muc-1 vaccine.
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | MUC1 Poly-ICLC
Number analyzed (Participants) | 39
participants | 39

3. Secondary Outcome: Number of Participants With Adverse Events Associated With the Study Agent
Description: Laboratory monitoring including Toxicity laboratory test or monitored through out the study up to week 54.
Time Frame: 54 weeks
Measure: Number; unit: participants
Arm/Group | MUC1 Poly-ICLC
Number analyzed (Participants) | 39
participants | 39

ADVERSE EVENTS:
Arm/Group | MUC1 Poly-ICLC
Serious Adverse Events (participants affected / at risk) | 0/39
Other Adverse Events (participants affected / at risk) | 39/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MUC1 Poly-ICLC (N=39)
injection site discomfort/ reddness (Skin and subcutaneous tissue disorders) | 39 (39)
Fatigue (Immune system disorders) | 3 (3)
Headache (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes